CLINICAL TRIAL: NCT03938714
Title: Hemorrhoidectomy in Patients With Grade III and IV Disease:Harmonic Scalpel Compared With Conventional Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Safia Zahir Ahmed, principal Investigator, Services Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB/503/SIMS
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Hemorrhoidectomy; Third Degree Hemorrhoids; Fourth Degree Hemorrhoids; Operative Time; Postoperative,Pain; Length of Stay
Keywords: VAS pain score; Harmonic Scalpel Hemorrhoidectomy; Conventional Hemorrhoidectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Hemorrhoidectomy

STUDY DESIGN:
Intervention Model Description: Coagulating Shears ® model
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CH( Conventional Hemorrhoidectomy) (Active Comparator): Closed Conventional Hemorrhoidectomy
  Interventions: Procedure: Hemorrhoidectomy
- HS( Harmonic Scalpel) (Experimental): Harmonic Scalpel Hemorrhoidectomy
  Interventions: Procedure: Hemorrhoidectomy

INTERVENTIONS:
Procedure: Hemorrhoidectomy — Excision of third and fourth degree hemorrhoids
  Other Names: Ferguson Closed Hemorrhoidectomy

SUMMARY:
Hemorrhoidectomy is the treatment of choice for grade 3 and 4th degree hemorrhoids. Various surgical technique has been used to improve the outcome of the procedures performed in respect to operative time ,post operative pain and hospital stay. This study compares the conventional closed technique with harmonic scalpel technique which is a device regulated with ultrasonic waves to perform the procedure with minimal postoperative complication as well as decreasing the prolong stay in hospital.

DETAILED DESCRIPTION:
INTRODUCTION:

Ferguson closed hemorrhoidectomy is conventional procedure in 3rd and 4th degree hemorrhoids but recent advances in harmonic scalpel have shown to produce favorable results. Comparison of these two is studied in terms of pain outcome as patient perceives, operative time and duration of hospital stay.

OBJECTIVES:

To compare the outcome of conventional hemorrhoidectomy versus harmonic scalpel in III and IV degree hemorrhoids.

STUDY DESIGN:

Randomized controlled trial

STUDY SETTING:

The study was conducted in surgical unit 1, Services hospital, Lahore.

DURATION OF STUDY:

Study was completed in six months after the approval of synopsis i.e. from 27th August 2015 to 26th February 2016.

DATA COLLECTION PROCEDURE:

After approval from hospital ethical committee, 100 patients fulfilling the inclusion criteria had been recruited from outdoor and emergency department. A detailed history had been taken including demographic data (age, address) and all patients had been clinically examined .Patients was divided in two groups randomly using random number tables. Group A: Conventional hemorrhoidectomy. Group B: harmonic scalpel hemorrhoidectomy. Patients had been requested to sign an informed consent. They had been assured regarding confidentiality and expertise used for the procedure. All procedures had been performed by a single surgical operating team to control bias. Per operatively operative time was noted. Post operatively pain had been assessed in 24 hours , mean hospital stay was measured in days from postoperative day till day of discharge (as per operational definition). All data had been collected and recorded on the attached Performa.

ELIGIBILITY:
Inclusion Criteria:

* Patients between age 20-60 years, both male and female with III and IV degree hemorrhoids diagnosed during last 1 year.

Exclusion Criteria:

* • Patients with permenantly prolapsed hemorrhoids limited to one quadrant only and had been assessed on per rectal examination and proctoscopy

  * Any other anorectal pathology such as anal fissure ,fistula or anal cancer on history and per rectal examination
  * Previous anal surgery assessed by history and per rectal examination
  * Inability to give informed consent
  * ASA grade III/IV on detailed history, clinical examination and laboratory findings e.g. deranged hepatic(AST/ALT >40IU/L) and renal profile ( creatinine >1:2mg/dl)and evidence of ischemic heart disease(annexure attached).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-08-27 (Actual); Primary Completion 2016-02-26 (Actual); Study Completion 2016-02-28 (Actual)

PRIMARY OUTCOMES:
Operative Time | The time was monitored from incision to the dressing approximately in 15 minutes to 50 minutes
  from start of incision to the dressing in minutes
post operative pain | Each Patient was measured in 24 hours
  On Visual analogue scale, a scale to measure pain and it ranges between 0-10. Scale 0-1 means no pain, 2-4 means mild pain,5-7 means moderate pain and 8-10 means severe pain. and it was measured post-operative in 24 hours
Hospital Stay | the Duration was measured from the day surgery performed till the day of Discharge i.e 1 to 5 days
  was measured in days from postoperative day till resolution of preoperative complaint of bleeding per rectum and VAS (<3)

CONTACTS AND LOCATIONS:
Overall Officials: Safia Z Ahmed, FCPS, Principal Investigator — Services Hospital
Locations (1):
- services Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
I want to share the abstract to other researches
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: data is available as the study is complete and for 12 month period
Access Criteria: will be shared upon request